CLINICAL TRIAL: NCT06729294
Title: Effect of Binaural Beat Music Played During Knee Arthroplasty With Spinal Anesthesia on Anxiety, Pain and Cortisol Levels.
Brief Title: Effect of Music Listened During Knee Arthroplasty With Spinal Anesthesia on Anxiety, Pain and Cortisol Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Fadime Ertural, Principal Investigator, Nuh Naci Yazgan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EBBMPDKASAAPC
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Spinal Anesthesia; Knee Arthroplasty
Keywords: binaural beat music; anxiety; pain; cortisol
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Binaural beat music is therapeutic music that provides auditory stimuli at different frequencies to each ear. However, the maximum sound levels of 60 dB help to relax and reduce stress. There are studies that show that a slower rhythm and a slower decibel music makes the heart beats compatible with the rhythm. Support from an audiologist will be sought to adjust the volume of the binaural beat music to 50 dB. Natural sounds such as birdsong, waterfalls, ocean, river and forest sounds will be added to the soothing components of the melodies, tones and rhythms embedded in the binaural beats and 60-minute music arrangements will be created in the computer program. The resulting binaural beat music will be loaded into the Goldplay GP-1001 brand Mp3 player and listened to using headphones.
  Interventions: Other: Binaural beat music recital
- Control group (No Intervention): Routine interventions will be applied to the control group without listening to music.

INTERVENTIONS:
Other: Binaural beat music recital — Binaural beats music is therapeutic music that provides auditory stimuli at different frequencies to each ear. However, the maximum sound levels are 60 dB, which helps to relax and reduce stress.
  Arms: Intervention group

SUMMARY:
The aim of this study is to examine the effects of binaural beat music played during spinal anesthesia knee arthroplasty on anxiety, pain and cortisol levels. The study was planned as a randomized controlled experimental design study. The hypotheses of the study are as follows;

* Binaural beat music played during spinal anesthesia knee arthroplasty has no effect on anxiety.
* Binaural beat music played during spinal anesthesia knee arthroplasty has an effect on anxiety.
* Binaural beat music played during spinal anesthesia knee arthroplasty has no effect on pain levels.
* Binaural beat music played during spinal anesthesia knee arthroplasty has an effect on pain levels.
* Binaural beat music played during spinal anesthesia knee arthroplasty has no effect on cortisol levels.
* Binaural beat music played during spinal anesthesia knee arthroplasty has an effect on cortisol levels.

A sample group will be formed with 20 patients in the intervention group and 20 patients in the control group. Binaural beat music will be played in the intervention group during the surgical procedure, and routine interventions will be applied to the control group.

Data collection in the intervention group is as follows;

* Patients will be interviewed in the surgery clinic before surgery and the descriptive characteristics form and the State Anxiety Inventory Form will be filled out.
* The 1st measurement of hemodynamic data will be recorded immediately before the surgery
* A musical concert will be started as soon as the surgery begins
* The musical concert will end when the surgery ends
* The 2nd measurement will be recorded immediately after the surgery ends
* In the post-surgery collection unit, the State Anxiety Inventory Form and the Visual Comparison Scale will be used, and a blood sample will be taken to determine cortisol values.

The control group data collection methods are as follows;

* Patients will be interviewed in the surgical clinic before surgery and the descriptive characteristics form and the State Anxiety Inventory Form will be filled in
* The first measurement of hemodynamic data will be recorded immediately before the surgical procedure
* The second measurement will be recorded immediately after the surgical procedure is completed
* Blood samples will be taken in the post-surgical recovery unit to determine the State Anxiety Inventory Form, Visual Comparison Scale and cortisol values.

DETAILED DESCRIPTION:
Knee arthroplasty is one of the most commonly used surgeries in orthopedics. Pain and anxiety are two main problems among patients undergoing orthopedic surgeries.

Being conscious during spinal anesthesia, potential risk, and expectation of postoperative pain contribute to anxiety and fear. Since the patient is fully conscious throughout the procedure, patients undergoing spinal anesthesia are more aware of the noise in the environment. Noise can cause stress, changes in the autonomic nervous system, and increase anxiety.

On the other hand, the surgical procedure itself also causes anxiety in the patient. Fear of surgical failure, lack of knowledge of the anesthesia methodology, possible risks of anesthesia, fear of the unknown, and expected pain during postoperative recovery cause increased anxiety.

The pain and anxiety experienced by surgical patients bring about psychological and physiological changes that significantly affect the course of the surgery, the recovery process, and the prognosis. Anxiety increases cortisol secretion through the autonomic nervous system. However, postoperative anxiety affects the pain response and strengthens the pain perception experienced by the patient. Since the intensity of pain can vary depending on the patient's anxiety, relieving anxiety can also facilitate pain management. Anxiety strengthens the perception of pain, and pain also causes anxiety in patients. In addition, anxiety and pain can reduce patient satisfaction. The irregularity in these psychological and physiological parameters caused by pain and anxiety can be reduced using pharmacological and non-pharmacological interventions. Music-based interventions are non-invasive, economical and non-pharmacological nursing interventions that do not require special skills to be applied, are safe, and also reduce pain and anxiety. Since they do not require a physician's order and have minimal fatal and ethical concerns, they can be easily incorporated into nursing care. Music-based interventions reduce pain and anxiety by distracting attention from stressful events such as pain and anxiety, allowing the music to focus on itself and related experiences/memories, i.e. another stimulus. The anxiolytic effect of music is achieved by suppressing the nervous system due to decreased adrenergic activity and neuromuscular stimulation. Music also stimulates the brain's limbic system to secrete endorphins, providing a sense of well-being. As a result, it reduces pain by increasing endorphin secretion and creating pleasant feelings. Music-based interventions can also reduce anxiety specifically by physiologically acting on the hypothalamic-pituitary-adrenal axis and reducing cortisol levels.

There is increasing interest in music interventions using binaural beats because it normalizes arrhythmias and provides relaxation in surgical patients. Binaural beat music is a therapeutic tool used to reduce anxiety and pain in patients undergoing surgical procedures. It has been reported that binaural beat music is successful as a non-pharmacological treatment method and is more effective than general music in reducing anxiety.

Music-based interventions for surgical pain and anxiety have been evaluated in many studies over the past few decades, but there are differences in the type and duration of intervention, the length of the evaluation, and other methodological issues. In this study, the intervention group will be provided with listening to music with headphones during the surgical procedure. Because therapeutic environments such as operating rooms are quiet, relatively secluded, and away from noise, which increases the success rate. However, in addition to the use of tools such as hammers, suction devices, and anesthetic monitors during orthopedic surgical procedures, the noise level associated with metal equipment also contributes to the noise level of operating rooms. While the noise level exceeds 100 dB more than 40% of the time in orthopedic surgical procedures, the highest noise level reached during the surgical procedure is over 120 dB. It has been stated that using headphones together with music to keep patients away from noise can reduce the anxiety caused by noise in the operating room and increase overall patient satisfaction. Using headphones increases a patient's focus on music and prevents other people nearby from being disturbed. Since patients receiving spinal anesthesia are more aware of the noise in the environment, in our study, the intervention group will be isolated from the noise by having them listen to music through headphones during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are older than 18 years,
* Who have undergone unilateral knee arthroplasty under spinal anesthesia for the first time,
* Who can communicate verbally,
* Who are in the ASA 1-2-3 group,
* Who do not have a neurological or psychiatric diagnosis will be included in the study.
* Since cortisol levels will be measured in our study, the first cases of the day will be included in the study.

Exclusion Criteria:

* Patients who refused to participate in the study were those with hearing impairment due to age or disease,
* Those who had any contraindications for spinal anesthesia,
* Those who were transferred to intensive care after the procedure,
* Those who developed complications during and after the procedure,
* Those who underwent general anesthesia,
* Those whose type of anesthesia was changed during surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory | Through study completion, an average of 2 months
  It is the State Anxiety Inventory Form that will be used for the subjective evaluation of patients' anxietyThe State Anxiety Inventory Form is a highly sensitive tool for assessing sudden changes in emotional reactions.
Visual Analog Scale | Through study completion, an average of 2 months
  The Visual Comparison Scale, which will be used to evaluate the level of pain and patient satisfaction with knee arthroplasty, consists of a 10 cm long horizontal line.
Cortisol level | Through study completion, an average of 2 months
  Anxiety increases cortisol secretion via the autonomic nervous system, causing an increase in cortisol levels. In this study, blood cortisol levels will be evaluated as objective data of anxiety.Cortisol levels gradually decrease throughout the day, exhibiting a 24-hour circadian rhythm. Cortisol levels are highest in the morning and lowest at midnight. To avoid being affected by this circadian shift, the first cases of the day will be included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Fadime Ertural, Principal Investigator — Nuh Naci Yazgan Üniversity; Salime Mucuk, Study Director — Erciyes Üniversty; Yeliz Sürme, Study Chair — Erciyes Üniversty; Gülden Küçükakça Çelik, Study Chair — Hacı Bektaş Veli Üniversty
Locations (1):
- Kayseri City Hospital, Kocasinan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I won't share it right now because it's a work in progress.